CLINICAL TRIAL: NCT02381275
Title: Baseline Characteristics and Long Term Clinical Outcomes of Patients Using Malawi's New First Line Antiretroviral Regimen at Lighthouse: The Lighthouse Tenofovir Cohort
Brief Title: The Lighthouse Tenofovir Cohort Study
Acronym: LighTen
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lighthouse Trust (Other)
Collaborators: Heidelberg University (Other); Ministry of Health, Malawi (Other Government); University of Cologne (Other)
Responsible Party: Principal Investigator, Sam Phiri, PhD, MSc, DCM, Executive Director, Lighthouse Trust
Other Study IDs: Lighten Cohort Study
Record Dates: First submitted 2015-02-24; First posted 2015-03-06 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Chronic Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Observe long-term outcomes of patients using Tenofovir based antiretroviral therapy at the Lighthouse Clinics

SUMMARY:
Lighthouse, in cooperation with the University Heidelberg Public Health Institute and the University Köln (Cologne) would like to set up a cohort to study baseline characteristics and long-term clinical outcomes of patients using Tenofovir based Antiretroviral Therapy at the Lighthouse. As of March 2014, patients above 18 years and giving informed consent coming to the Lighthouse to newly initiate ART will be approached to enroll in the cohort.

The results will be disseminated both nationally at the Ministry of Health Technical Working Group (TWG), at the annual Research Dissemination and Best Practices conferences of the College of Medicine and National AIDS Commission as well as internationally. The results will also be written up for publication in appropriate peer-reviewed journals.

DETAILED DESCRIPTION:
The proposed observational cohort study will lead to improved identification of patients with virological failure and adverse drug effects, improved identification of relevant co-morbidities and result in better individual management. More importantly however, the results will allow estimates for the proportion of the described complications in the overall Malawian treatment cohort. This claim can be exemplified by the retrospective analysis of patients at the Lighthouse who were switched from the new 5A regimen to 6 A regimen as a result of adverse effects of Efavirenz.

The aim of this study is to describe baseline clinical characteristics and long-term outcomes of patients using Tenofovir based antiretroviral therapy at the Lighthouse Clinics. The specific objectives are outlined below:

Objective 1: To determine the prevalence of renal dysfunction at enrolment and during follow-up among adult HIV-infected individuals starting ART.

Objective 2: To determine the prevalence of Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infections among adult HIV-infected individuals starting ART and during treatment follow-up.

Objective 3: To determine the prevalence of non-communicable co-morbidities during treatment follow-up of HIV-infected individuals starting ARTand during treatment follow-up.

The study will take place at the Lighthouse, a tertiary referral ART centre, with over 25,000 patients, in Lilongwe, Malawi. Considering the study cost and power to detect a prevalence of 22% for renal impairment, we expect to have a convenience sample size of at least 850 patients at the end of three year follow-up period. The current retention at three years is almost 56%. Using this retention, we will therefore enrol almost 1,500 patients starting ART.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able and willing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients initiating Tenofovir based ART regimen at the Lighthouse clinics
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV-infected individuals with renal dysfunction | 36 months post ART initiation
  Patients will be followed in the clinic up to 36 months

SECONDARY OUTCOMES:
Proportion of HIV-infected individuals with HIV/ HBV and HCV infections | 36 months post ART initiation
  Patients will be followed in the clinic up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Lighthouse Clinic, Lilongwe, Malawi

REFERENCES:
- [Derived] Steffen HM, Viola E, Thawani A, Kachere LG, Huwa J, Wallrauch C, Kasper P, Neuhann F, Heller T, Winkler V, Rambiki E, Mahanani MR. Blood pressure, weight change and incident hypertension after switching to dolutegravir in treatment-experienced people living with HIV. AIDS. 2025 Jul 24. doi: 10.1097/QAD.0000000000004309. Online ahead of print. PMID 40704988
- [Derived] Steffen HM, Mahanani MR, Neuhann F, Nhlema A, Kasper P, de Forest A, Chaweza T, Tweya H, Heller T, Chiwoko J, Winkler V, Phiri S. Blood pressure changes during tenofovir-based antiretroviral therapy among people living with HIV in Lilongwe, Malawi: results from the prospective LighTen Cohort Study. Clin Res Cardiol. 2023 Nov;112(11):1650-1663. doi: 10.1007/s00392-023-02253-w. Epub 2023 Jul 6. PMID 37414923
- [Derived] Kasper P, Nhlema A, de Forest A, Tweya H, Chaweza T, Mwagomba BM, Mula AM, Chiwoko J, Neuhann F, Phiri S, Steffen HM. 24-h-Ambulatory Blood Pressure Monitoring in Sub-Saharan Africa: Hypertension Phenotypes and Dipping Patterns in Malawian HIV+ Patients on Antiretroviral Therapy. Glob Heart. 2021 Oct 13;16(1):67. doi: 10.5334/gh.945. eCollection 2021. PMID 34692392